CLINICAL TRIAL: NCT04854616
Title: Cessation of Smoking Trial in the Emergency Department
Acronym: CoSTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R208399; NIHR129438 (Other Grant/Funding Number: NIHR HTA (UK))
Record Dates: First submitted 2021-03-26; First posted 2021-04-22 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation; Electronic Cigarette Use; E-Cig Use; Vaping
Keywords: intervention; emergency department; e-cigarette; electronic cigarette; A&E; Accident and Emergency; vaping; behavioural intervention; stop smoking services
MeSH Terms: conditions — Smoking Cessation; Vaping; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoSTED Intervention (Experimental): CoSTED is an opportunistic smoking cessation intervention comprising three elements:
  1. brief smoking cessation advice
  2. the provision of an electronic cigarette (e-cigarette) and training in its use
  3. referral to stop-smoking services
  Interventions: Behavioral: CoSTED Intervention
- Treatment as Usual (No Intervention): Signposting to NHS smoking cessation services through provision of written information about local services.

INTERVENTIONS:
Behavioral: CoSTED Intervention — Brief smoking cessation advice, the provision of an e-cigarette starter kit and training in its use, and referral to stop smoking services.
  Arms: CoSTED Intervention

SUMMARY:
The Cessation of Smoking Trial in the Emergency Department (CoSTED) is an National Institute for Health Research (NIHR) Health Technology Assessment (HTA) funded randomised controlled trial (RCT). The research question is "in people attending the Emergency Department who smoke, does a brief intervention (including the provision of an electronic cigarette (e-cigarette) and referral to stop smoking services) increase smoking cessation in comparison with usual care and is it cost effective?" The trial includes an internal pilot, health economic evaluation and process evaluation. The primary outcome is smoking cessation, self-reported as continuous smoking abstinence, biochemically validated by carbon monoxide monitoring with cut off of ≥8ppm. The sample size is 972 (486 in intervention and control) across 6 sites.

DETAILED DESCRIPTION:
Research question:

In people attending the Emergency Department who smoke, does a brief intervention (including the provision of an e-cigarette and referral to stop smoking services) increase smoking cessation in comparison with usual care and is it cost effective?

Background:

Tobacco smoking is the leading cause of years of life lost in the United Kingdom (UK), and negatively impacts significantly on physical health conditions and recovery outcomes from injury or surgery. Currently, smoking prevalence is recorded at approximately 15% of the population, but this masks substantial variation between different population groups. Patient and Public Involvement (PPI) development work demonstrates that prevalence of smoking for people attending the emergency department is approximately 24%. Most current smokers will, if asked, state that they want to quit, but need support. The National Health Service (NHS) long term plan and the Tobacco control plan for England recommend smokers are supported to quit at every contact with the health service by 2023/4. To date there have been no RCTs of smoking cessation support in the Emergency Department (ED) setting in the UK, which potentially provides a highly motivating opportunistic route to intervention.

Aims and objectives:

To undertake an RCT, with internal pilot, comparing a brief intervention (including provision of an e-cigarette and referral to local smoking cessation services), assessing long term smoking abstinence, in people attending Emergency Departments.

1. To run an internal pilot study, with clear stop/go criteria, primarily to test recruitment systems
2. To definitively test real-world effectiveness of an ED based smoking cessation intervention in comparison with usual care, by comparing smoking abstinence at 6 month follow-up between trial groups
3. To undertake a cost effectiveness analysis of the intervention in comparison with usual care, from an NHS and personal social services (PSS) perspective
4. To undertake an embedded mixed-methods process evaluation to assess delivery, implementation, fidelity and contamination

Methods:

Randomised Controlled Trial of people who smoke attending an Emergency Department, with an internal pilot, health economic evaluation and process evaluation. The primary outcome is smoking cessation, self-reported as continuous smoking abstinence, biochemically validated by carbon monoxide monitoring with cut off of ≥8ppm. The sample size is 972 (with a power of 90% and a difference in quit rates between the groups of 6%).

Anticipated impact and dissemination:

The investigators will definitively test an ED based smoking cessation intervention and make recommendations for future implementation if effective. The intervention has the potential to reduce smoking prevalence by at least 6% based on existing evidence, impacting on improved long term health outcomes for approximately 334,000 members of the UK population if adopted across the NHS. Results will be disseminated at international conferences and published in leading journals to reach academic experts, through NHS networks and the Royal College of Emergency Medicine to reach commissioners, managers and members of the public.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old who are current daily tobacco smokers
2. Current daily tobacco smoker (self-reporting smoking of at least one cigarette per day)
3. Attending the ED for medical treatment (or accompanying a patient attending for medical treatment)
4. Submitting an expired carbon monoxide (CO) breath test reading of more than ≥8 parts per million (ppm).

Exclusion Criteria:

1. Requiring immediate medical treatment as defined by the treating clinician.
2. In police custody.
3. Known history of allergy to nicotine replacement products.
4. Currently defined as dual users - already using an e-cigarette daily as well as smoking conventional cigarettes.
5. Without the capacity to give informed consent for participation in the study
6. Have taken part in the CoSTED trial already

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Continuous smoking abstinence | 6 months after randomisation
  The primary outcome is smoking cessation, self-reported as continuous smoking abstinence, biochemically validated by carbon monoxide monitoring with cut off of ≥8ppm.This is according to the Russell standard, stated as: continuous abstinence (Russell Standard) [ Time Frame: Six months post quit date ] Self-report of smoking not more than five cigarettes from the Quit date, supported by biochemical validation (expired air carbon monoxide)

SECONDARY OUTCOMES:
7-day point prevalence abstinence | 6 months after randomisation
  7-day point prevalence abstinence, i.e. current smoking status, Self-report of having smoked no cigarettes (not even a puff) in the past seven days, biochemically validated by carbon monoxide monitoring with cut off of ≥8ppm
Number of quit attempts | Baseline and 6 months after randomisation
  Numerical value
Time to relapse (if applicable) | 6 months after randomisation
  (if applicable)
Number of cigarettes per day | Baseline and 6 months after randomisation
  Numerical value
Nicotine dependence | Baseline and 6 months after randomisation
  At baseline & 6 month follow up, participants will be asked about their nicotine dependence using the Fagerstrom test for nicotine dependence
Number of times using an e-cigarette per day | Baseline and 6 months after randomisation
  Numerical value
Self-reported dry cough or mouth or throat irritation | Baseline and 6 months after randomisation
  This will be measures as a yes/no response for symptoms in the last week
Motivation to stop smoking | Baseline and 6 months after randomisation
  Motivation to Stop Smoking scale (MTSS)
Self-reported use of healthcare services in the last 3 months | Baseline and 6 months after randomisation
  At baseline & 6 month follow up, participants will be asked about their use of GP services in the past 3 months including number of times they have attended face-to-face and telephone appointments
Self-reported use of smoking cessation services in the last 3 months | Baseline and 6 months after randomisation
  At baseline & 6 month follow up, participants will be asked about their use of smoking cessation services in the past 3 months and number of times attended
Quality of Life questionnaire | Baseline and 6 months after randomisation
  At 6-month follow-up, quality of life will be assessed using EQ-5D-5L where a higher value equates to a lower quality of life (i,e. worse outcome)
Adverse events | 1, 3, and 6 months after randomisation
Smoking status | 1, 3 & 6 months after randomisation
  This is the only outcome that will be asked at 1-month, 3-months and 6-months from randomisation. This will be a binary question of "have you smoked even a single puff of a cigarette in the past 2 weeks"- point prevalence abstinence
Frequency of e-cigarette use in the past 6 months | 6 months after randomisation
  E-cigarette usage in the past 6 months
Long term follow-up 7-day point prevalence abstinence | Measured between 12 and 18 months post randomisation
  7-day point prevalence abstinence, i.e. current smoking status, Self-report of having smoked no cigarettes in the past seven days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Pope, MD, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data underlying the main trial results will be available in a public, open access repository immediately following publication of the major findings of the study. Details of the repository and a persistent URL will be provided on publication of the main results. Study protocol, statistical analysis plan, informed consent form, and other documents will also be available.

REFERENCES:
- [Background] Notley C, Clark L, Belderson P, Ward E, Clark AB, Parrott S, Agrawal S, Bloom BM, Boyle AA, Morris G, Gray A, Coats T, Man MS, Bauld L, Holland R, Pope I. Cessation of smoking trial in the emergency department (CoSTED): protocol for a multicentre randomised controlled trial. BMJ Open. 2023 Jan 18;13(1):e064585. doi: 10.1136/bmjopen-2022-064585. PMID 36657751
- [Derived] Ward E, Belderson P, Clark A, Stirling S, Clark L, Pope I, Notley C. How do people quit smoking using e-cigarettes? A mixed-methods exploration of participant smoking pathways following receiving an opportunistic e-cigarette-based smoking cessation intervention. Addiction. 2024 Dec;119(12):2185-2196. doi: 10.1111/add.16633. Epub 2024 Sep 10. PMID 39252616
- [Derived] Pope I, Clark LV, Clark A, Ward E, Belderson P, Stirling S, Parrott S, Li J, Coats T, Bauld L, Holland R, Gentry S, Agrawal S, Bloom BM, Boyle AA, Gray AJ, Morris MG, Livingstone-Banks J, Notley C. Cessation of Smoking Trial in the Emergency Department (COSTED): a multicentre randomised controlled trial. Emerg Med J. 2024 Apr 22;41(5):276-282. doi: 10.1136/emermed-2023-213824. PMID 38531658
- [Derived] Belderson P, Ward E, Pope I, Notley C. Selecting an e-cigarette for use in smoking cessation interventions and healthcare services: findings from patient and public consultation for the COSTED trial. BMJ Open. 2024 Mar 4;14(3):e078677. doi: 10.1136/bmjopen-2023-078677. PMID 38443079
- See also: CoSTED trial web page — https://pubmed.ncbi.nlm.nih.gov/36657751/